CLINICAL TRIAL: NCT07309120
Title: Nutrition Ameliorates the Muscle Loss of Pre-sarcopenia in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202100551A3
Record Dates: First submitted 2025-11-18; First posted 2025-12-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Low Muscle Mass; Low Muscle Strength; Low Physical Function
Keywords: metabolomics; supplemenation; pre-sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protein Supplementation Group (Experimental)
  Interventions: Dietary Supplement: Participants consume two sachets daily over a 12-week intervention period.

INTERVENTIONS:
Dietary Supplement: Participants consume two sachets daily over a 12-week intervention period. — Each 8 g serving provided 35 kcal, comprising 4.1 g of protein, 1 g of fat, and 2.4 g of carbohydrates.

SUMMARY:
This study evaluates the effects of a 12-week leucine-enriched protein supplementation in adults aged 60 years and more. Participants will undergo assessments of muscle mass and function, as well as metabolic profiles in blood, urine, and feces before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent.
2. Participants who attend health check-ups at Songshan District, Taipei City, or at the Wellness Cultural Village, or who have participated in the pilot study.
3. Adults aged 60 years or older, male or female.
4. Able to ambulate independently.
5. Meets at least one of the following sarcopenia criteria:

Grip strength: Men < 28 kg; Women < 18 kg Gait speed: < 1.0 m/s Muscle mass (appendicular skeletal muscle mass / height²): Men < 7.0 kg/m²; Women < 5.7 kg/m²

Exclusion Criteria:

1. Impaired renal function.
2. Allergy or intolerance to protein supplements.
3. Currently undergoing cancer treatment.
4. Autoimmune diseases.
5. Assessed by a physician as unsuitable to participate.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Appendicular Skeletal Muscle Index (ASMI) | Baseline and 12 weeks after intervention
  Muscle mass was assessed using bioelectrical impedance analysis (Tanita MC-780MA). The appendicular skeletal muscle index (ASMI, kg/m2) was calculated as appendicular skeletal muscle mass (ASM, kg) divided by height squared (m²).
Handgrip Strength (HGS) | Baseline and 12 weeks after intervention
  Functional performance was evaluated by handgrip strength (HGS, kg), measured with a digital hand dynamometer.
Gait speed (m/s) | Baseline and 12 weeks after intervention
  Gait speed was assessed as the time required to walk a 4 meters, expressed in meters per second (m/s).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Guishan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Due to ethical and privacy considerations, individual participant data will not be publicly available. De-identified data may be shared upon reasonable request and with approval from the institutional review board.

REFERENCES:
- [Background] Prado CM, Landi F, Chew STH, Atherton PJ, Molinger J, Ruck T, Gonzalez MC. Advances in muscle health and nutrition: A toolkit for healthcare professionals. Clin Nutr. 2022 Oct;41(10):2244-2263. doi: 10.1016/j.clnu.2022.07.041. Epub 2022 Aug 7. PMID 36081299
- [Background] Lee SY, Lee HJ, Lim JY. Effects of leucine-rich protein supplements in older adults with sarcopenia: A systematic review and meta-analysis of randomized controlled trials. Arch Gerontol Geriatr. 2022 Sep-Oct;102:104758. doi: 10.1016/j.archger.2022.104758. Epub 2022 Jun 24. PMID 35777246

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT07309120/Prot_SAP_000.pdf